CLINICAL TRIAL: NCT07254962
Title: CApecitabine Prior to TUmor Resection in Ent Oncology (CAPTURE)
Acronym: CAPTURE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Marco Mascarella, Principal Investigator, Clinical professor, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-37-2026-12048
Record Dates: First submitted 2025-11-16; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Head Neck Cancer; Mouth Cancer; Throat Cancer; Larynx Cancer; Skin Cancer Face
Keywords: window of opportunity; surgery; neoadjuvant; capecitabine; Head and neck cancer; HPV-negative
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Laryngeal Neoplasms | interventions — Capecitabine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Patients will receive standard of care surgery (no intervention prior to surgery)
  Interventions: Other: Standard of Care (SOC)
- Capecitabine (Experimental): Patients will receive capecitabine prior to surgery
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Patients will receive fixed-dose capecitabine prior to surgery
  Arms: Capecitabine
Other: Standard of Care (SOC) — Standard of care (no intervention until surgery)
  Arms: Standard of Care

SUMMARY:
head and neck squamous cell carcinoma (HNSCC) is a type of cancer that affects areas such as the mouth, throat, and voice box. Despite medical progress, little has changed in the care for patients with HPV-negative cancer. The standard care involves surgery followed by radiation or chemotherapy if needed. However, delays in starting treatment - especially beyond six weeks - are linked to worse outcomes. Many patients also experience cancer returning within two years, often making it harder to treat. This study aims to improve outcomes by giving patients a short course of capecitabine, a chemotherapy pill, before surgery. Capecitabine is easier to tolerate than traditional intravenous chemotherapy and has shown promising results in shrinking tumors. Researchers believe that starting this oral treatment early could reduce delays, shrink tumors, make surgery less complex, and improve survival. The clinical trial will randomly assign patients with newly diagnosed stage III or IVa HPV-negative head and neck cancer to receive either standard care or capecitabine before surgery. Surgery will be performed within six weeks of diagnosis, followed by additional therapy as needed. The study will measure how well the tumor responds under the microscope after surgery, how much it shrinks on scans, the safety of the treatment, and cancer-free survival at two years. It will also explore biological markers linked to treatment response.

If successful, this approach could offer a simpler, faster, and more effective way to treat head and neck cancer, leading to earlier treatment, less invasive surgery, and improved patient outcomes. The study plans to include about 62 patients to evaluate the benefits of this new treatment strategy

ELIGIBILITY:
Inclusion Criteria:

* • Previously untreated, histologically confirmed non-HPV related HNSCC and radiologically or histologically confirmed stage I or IVA (AJCC 8th edition).

  * No evidence of distant metastatic disease.
  * Able to undergo protocol therapy, including necessary imaging and surgery.
  * If female: may participate if not actively pregnancy nor breastfeeding.
  * If male: must agree to refrain from donating sperm and must either be abstinent or agree to use contraception.
  * Performance status (ECOG) of 0, 1 or 2.

Exclusion Criteria:

* History of immunodeficiency, HBV, HCV, HIV. No HBV, HCV or HIV testing is required unless mandated by local health authority.
* Active infection requiring systemic therapy.
* Previous allogenic tissue/solid organ transplant.
* Known severe hypersensitivity (≥ Grade 3) to capecitabine, its active substance and/or any of its excipients.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Known DYPD mutation.
* Known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the trial.
* Received prior systemic anticancer therapy including investigational agents for the current malignancy prior to allocation.
* Currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of trial treatment.
* Known additional malignancy that is progressing or requires active treatment within the past (5 years), excluding basal cell carcinoma or cutaneous squamous cell carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic response | From initiation of capecitabine to surgery
  modified Ryan criteria: score based on the following: no viable cancer, rare groups of cancer cells, residual cancer with tumor regression, no evident tumor regression

SECONDARY OUTCOMES:
Treatment toxicity (grade 3 or greater) | Within first 60 days of treatment initiation
  CTCAE version 5 grade 3 or greater

OTHER OUTCOMES:
Disease-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Disease-Free Survival: length of time after definitive therapy during which free from cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mascarella, MD, MSc, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre

IPD SHARING:
Plan to Share IPD: Undecided